CLINICAL TRIAL: NCT02992782
Title: Decongestive Progressive Resistance Exercise With Advanced Compression for Breast Cancer Related Lymphedema Management (DREAM): A Pilot Randomized Control Trial
Brief Title: Decongestive Exercise and Compression for Breast Cancer Related Lymphedema Management
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA - CC 16-1026
Record Dates: First submitted 2016-12-10; First posted 2016-12-14 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasm; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Standard of Care; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (Active Comparator): Standard care Intervention: including a home program of therapeutic (decongestive) exercise, which will include active, non-resistive motion of the involved limb. Participants will perform the exercise once daily for about 10 minutes and will be required to wear their compression sleeve for at least 12 hours per day, each day of the week. After 24 weeks, they will be given the opportunity to take part in the decongestive progressive resistance exercise program and will be provided with an adjustable compression garment to use during exercise.
  Interventions: Behavioral: Standard Care
- Exercise and Compression Garment (Experimental): Intervention will include having participants wear a compression sleeve during exercise. They will wear the sleeve while carrying out the decongestive progressive resistance exercise program and will continue wearing their day-time compression garment for at least 12 hours per day, each day of the week. They will attend a supervised decongestive progressive resistance exercise program twice a week for 12 weeks at the Cancer Rehabilitation Clinic in Corbett Hall at the University of Alberta. Exercise session will take approximately 60-90 minutes. After 12 Weeks, participants will continue the same program twice weekly for an additional 12 weeks in a community-based fitness center or at home.
  Interventions: Behavioral: Exercise and Compression Garment
- Exercise and Adjustable Compression Wrap (Experimental): Intervention will include having participants will be fitted for an adjustable compression wrap. They will be required to wear the adjustable compression wrap during the decongestive progressive resistance exercise program and will continue wearing their compression sleeve at least 12 hours per day, each day of the week. They will attend a supervised decongestive progressive resistance exercise program twice a week for 12 weeks at the Cancer Rehabilitation Clinic in Corbett Hall at the University of Alberta. Exercise session will take approximately 60-90 minutes. After 12 weeks, participants will continue the same program twice weekly for an additional 12 weeks in a community-based fitness centre or at home.
  Interventions: Behavioral: Exercise and Adjustable Compression Wrap

INTERVENTIONS:
Behavioral: Standard Care — Home program of decongestive exercise and daily use of a compression sleeve
  Arms: Standard Care
Behavioral: Exercise and Compression Garment — Decongestive progressive resistance exercise using flat-knit garment and daily use of a compression sleeve
  Arms: Exercise and Compression Garment
Behavioral: Exercise and Adjustable Compression Wrap — Decongestive progressive resistance exercise using adjustable compression wrap and daily use of a compression sleeve
  Arms: Exercise and Adjustable Compression Wrap

SUMMARY:
Women who have undergone breast cancer surgery may develop swelling of the arm on the side the breast cancer occurred. If the swelling becomes chronic it is called lymphedema. This study will examine the effect of a 12-week decongestive progressive resistance exercise with advanced compression on breast cancer related lymphedema. Our objective is to determine if breast cancer survivors are willing and able to wear advanced compression while exercising and if the combination will help to reduce their lymphedema. Twenty-four breast cancer survivors from Edmonton, Alberta will be enrolled in the one-year long study.

DETAILED DESCRIPTION:
Lymphedema is a swelling in the arm, chest wall and breast on the side of the breast cancer. Arm lymphedema develops as a result of breast cancer surgery and/ or radiation therapy. Compression therapy and exercise are commonly prescribed treatment to help reduce the arm swelling and to maintain the result. The exercise that is usually prescribed for lymphedema is called decongestive remedial exercise. It involves active, non-resisted movements that follow a specific order from proximal to distal and back proximally. The exercises start at the neck, move to the chest wall and then down the arm, and back.

Two different types of compression garments have been proposed to help reduce swelling when women are exercising. One compression garment is made with a stiffer, less elastic type of material and is called a "flat-knit" garment. The other garment, the "Adjustable Compression Wrap" is a garment with an adjustable elastic strapping system that helps to reinforce the compression on the arm. Recent research suggests that these specialized garments enhance the muscle pump effect on lymph flow; however, no research has been conducted to test whether this actually results in improvements in arm lymphedema volume.

Resistance exercise training helps to improve arm flexibility, strength, function, and quality of life in breast cancer survivors. Recent evidence has shown that breast cancer survivors with lymphedema, can safely perform resistance training (strength training), however, there is no impact (better or worse) on arm lymphedema volume.

To date, no studies have been performed combining all potential therapeutic approaches for lymphedema management: resistance exercise, a therapeutic decongestive exercise sequence, and compression therapy. Women in the experimental arms of this study will wear a compression garment when performing progressive resistance exercise that follows the decongestive sequence. We will examine the effect of the combined intervention on arm lymphedema volume, function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Is a female with a history of breast cancer;
2. Has undergone surgery, including sentinel lymph node biopsy or axillary lymph node dissection;
3. Has unilateral mild to moderate lymphedema of at least 200 ml or 10% inter-limb volume difference or a maximum of 40% and/or minimal volume difference of 100 ml or 5% in hand and forearm region;
4. Has chronic lymphedema, defined as lymphedema that has been present for at least 3 months;
5. Is in the lymphedema maintenance phase of conservative treatment;
6. Uses a well fitted compression sleeve (not older than 1 month) and is agreeable to wear the sleeve for a minimum of 12 hours per day (providing a minimum of 30 mm Hg of pressure);
7. Is agreeable to discontinuing other lymphedema treatments, including manual lymph drainage and intermittent pneumatic compression during the supervised intervention period of the study

Exclusion Criteria:

1. Are undergoing or are scheduled for chemotherapy, radiotherapy or biological therapy;
2. Present with limb infection, deep vein thrombosis, cellulitis, or have active metastatic disease;
3. Have any neurological, cognitive deficit or other uncontrolled health condition that may interfere with assessment and/or the progressive resistance exercise training intervention;
4. Have any contraindications related to wearing compression on the limb, including arterial insufficiency or congestive heart failure;
5. Have a body mass index (BMI) greater than 40 kg/m2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Arm Lymphedema Volume | Change from baseline to 12 weeks
  Lymphedema will be objectively measured using the Perometer (Pero-systems, Wipputal, Germany)

SECONDARY OUTCOMES:
Bioimpedance Analysis | Change from baseline to 12 weeks
  Bioimpedance analysis (BIA) will be used to assess extracellular fluid status within the arm
Upper body strength | Change baseline to 12 weeks
  One repetition maximum strength for bench press and seated row
Lower body strength | Change baseline to 12 weeks
  One repetition maximum strength for leg press
Shoulder range of motion | Change baseline to 12 weeks
  Range of motion measured with goniometer: forward flexion, abduction, external, internal and horizontal abduction movements
Lymphedema International Classification of Functioning (LYMPH-ICF) | Change baseline to 12-weeks
  Lymphedema-specific quality of life
Rand Short-form (SF): 36 | Change baseline to 12-weeks
  General health-related quality of life
Godin Leisure-time Questionnaire | Change baseline to 12-weeks
  Physical activity level in previous 4-week period
Body composition | Change baseline to 12-weeks
  Body mass index as calculated by body weight and height metrics
Body Image | Change baseline to 12-weeks
  Body Image and Relationship in past month
Tissue Composition | Change baseline to 12-weeks
  Magnetic Resonance Imaging: fat, water and muscle mass

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L McNeely, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
On completion of the study, data will be made available through the University of Alberta Libraries Dataserve Network
Time Frame: Not determined
Access Criteria: Pending